CLINICAL TRIAL: NCT01780155
Title: Candidate Genes Associated With Susceptibility to Bronchopulmonary Dysplasia and Retinopathy of Prematurity
Brief Title: Genes Associated With Bronchopulmonary Dysplasia and Retinopathy of Prematurity
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913031; 13-E-N031
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2019-08

CONDITIONS: Bronchopulmonary Dysplasia; Retinopathy of Prematurity; Prematurity; Pulmonary Disease
Keywords: Oxidative Stress; Hyperoxia; Brochopulmonary Dysplasia; Retinopathy of Prematurity; Very Low Birth Rate
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Retinopathy of Prematurity; Premature Birth; Lung Diseases; Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Parents and premature newborns with a birth weight less than or equal to1250 g from member institutions of the hospital network will be invited to participate in this study.

SUMMARY:
Background:

- Some premature babies develop bronchopulmonary dysplasia (BPD) and retinopathy of prematurity (ROP). BPD and ROP are long-term chronic diseases of the lungs and eyes, respectively. BPD is associated with receiving mechanical ventilation to treat respiratory distress syndrome, and causes lung inflammation and scarring. ROP is caused by poor development of blood vessels in the eyes, and may lead to blindness. Because not all premature babies develop BPD or ROP, researchers want to study the genes that could be associated with these diseases. They will look at both premature infants and their parents to see if there is a genetic component to BPD and ROP.

Objectives:

- To study genes that may be associated with BPD and ROP.

Eligibility:

* Premature babies born with a weight less than or equal to 1,250 grams.
* Parents of the premature babies.

Design:

* Parents will answer questions about the mother s health and pregnancy.
* Delivery and medical information will be collected during the baby s hospitalization for the first month after birth.
* Parents will provide a saliva sample from the inside of the cheek.
* A saliva sample will also be collected from the baby within 28 days of birth. If the baby needs tracheal aspiration (removal of fluid from the throat), tracheal fluid samples will also be collected.
* Parents will have followup interviews about their child s health 6 months, 12 months, and yearly for up to 6 years after birth.
* This is a genetic study only. Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Understanding the role of susceptibility genes for risk of BPD and ROP may lead to immediate identification of populations who require personalized medical care, and to the assessment of innovative prophylactic and therapeutic interventions in the future. Our purpose is to establish in our hospital network a prospective cohort of triads composed of premature newborns with a birth weight less than or equal to 1250 g and their parents, to examine the role of candidate susceptibility genes in the development of BPD and ROP. Our hypothesis is that the presence of single-nucleotide polymorphisms in candidate genes is associated with differential susceptibility to BPD and ROP. As an initial model, a loss-of-function substitution at position -617 of the NRF2 promoter region is hypothesized to be associated with a greater risk of severe BPD and prethreshold ROP in premature infants with a birth weight less than or equal to 1250 g.

ELIGIBILITY:
* INCLUSION CRITERIA:

Premature newborns with a birth weight less than or equal to 1250 g and their parents from the participating institutions that comprise the Fundacion Infant hospital network will be enrolled in this study after signing the informed consent.

EXCLUSION CRITERIA:

Premature newborns with a birth weight less than or equal to 1250 g with cyanotic congenital heart disease, congenital anomalies of the respiratory tract (for example, tracheoesophageal fistula, pulmonary hypoplasia, diaphragmatic hernia), eye malformations, or congenital immunodeficiencies. Newborns from parents (mother and/or father) who used in vitro fertilization products from donor banks will also be excluded from participating in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited irrespective of gender, ethnicity, race, or socio-economic status. Parents and premature newborns with a birth weight less than or equal to1250 g from member institutions of the hospital network will be invited to participate in this study.@@@
Sampling Method: Non-Probability Sample
Enrollment: 1068 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia; retinopathy of prematurity | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Kleeberger, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (8):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States
- Argentina (7):
  - Clinica Y Maternidad, Buenos Aires
  - Fundacion Infant, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto Medico de Obstretricia (IMO), Buenos Aires
  - Sanatario de los Arcos, Buenos Aires
  - Sanatorio de la Trinidad, Buenos Aires
  - Sanatorio Otamendi y Miroli, Buenos Aires

REFERENCES:
- [Background] Anderson CG, Benitz WE, Madan A. Retinopathy of prematurity and pulse oximetry: a national survey of recent practices. J Perinatol. 2004 Mar;24(3):164-8. doi: 10.1038/sj.jp.7211067. PMID 14999216
- [Background] Asikainen TM, Huang TT, Taskinen E, Levonen AL, Carlson E, Lapatto R, Epstein CJ, Raivio KO. Increased sensitivity of homozygous Sod2 mutant mice to oxygen toxicity. Free Radic Biol Med. 2002 Jan 15;32(2):175-86. doi: 10.1016/s0891-5849(01)00776-6. PMID 11796207
- [Background] Clyman R. Oxygen-saturation targets and outcomes in extremely preterm infants. J Pediatr. 2004 Mar;144(3):408. No abstract available. PMID 15032225